CLINICAL TRIAL: NCT03982992
Title: Phase 2 Study Evaluating the Safety, Tolerability and Efficacy of Allogeneic Donor Lymphocyte Infusions Combined With Blinatumomab in Patients With Treatment-Resistant Mixed Chimerism or Minimal Residual Disease of B-precursor Acute Lymphoblastic Leukemia After Allogeneic Stem Cell Transplantation
Brief Title: Allogeneic Donor Lymphocyte Infusions Combined With Blinatumomab
Acronym: DLI-TARGET
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of potential study subjects due to a change of standard of care treatment outside of clinical trials.
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Christian Schmidt, MD, Deputy Principal Investigator, Ludwig-Maximilians - University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-002314-31
Record Dates: First submitted 2019-06-03; First posted 2019-06-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: B Cell Precursor Acute Lymphoblastic Leukemia With Mixed Chimerism or Minimal Residual Disease After Allogeneic Stem Cell Transplantation; B-Cell Acute Lymphoblastic Leukemia; Acute Lymphoblastic Leukemia; Acute Lymphoblastic Leukemia in Remission; Acute Lymphoblastic Leukemia, Adult
Keywords: donor lymphocyte infusion; blinatumomab; combinatorial; minimal residual disease; MRD; mixed chimerism; MC; DLI-TARGET; acute lymphoblastic leukemia
MeSH Terms: conditions — Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DLI-TARGET (Experimental): 14d screening period: methotrexate, cytarabine, dexamethasone infusion i.th.
  Cycle 1 (all patients): d1-28: blinatumomab continuous infusion i.v., d4: allogeneic donor lymphocyte single infusion i.v., d29: methotrexate, cytarabine, dexamethasone infusion i.th.
  Cycle 2 (only patients with toxicity ≤ grade 2 CTCAE in cycle 1): d43-d70: blinatumomab continuous infusion i.v., d46: allogeneic donor lymphocyte single infusion i.v., d71: methotrexate, cytarabine, dexamethasone infusion i.th.
  Interventions: Drug: Blinatumomab in combination with donor lymphocyte infusion

INTERVENTIONS:
Drug: Blinatumomab in combination with donor lymphocyte infusion — Continuous blinatumomab infusion in combination with allogeneic donor lymphocyte infusion

SUMMARY:
This phase 2 study is designed to evaluate the safety, tolerability and efficacy of allogeneic donor lymphocyte infusions (DLI) combined with the bispecific T cell engager blinatumomab in B-precursor ALL patients who have mixed chimerism (MC) or are MRD-positive after allogeneic SCT and are refractory to at least one MRD- or MC-targeted therapy (i.e. blinatumomab, DLI, tyrosine kinase inhibitors or other agents).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with CD19+ B-precursor ALL (as determined by immunophenotyping) in hCR (defined as having less than 5% blasts in bone marrow) after allogeneic SCT.
2. One, or a combination of the following documented after an interval of at least 2 weeks since cessation of the most recent leukemia-targeting therapy (i.e. chemotherapy, immunotherapy or cellular therapy, except for intrathecal prophylaxis):

   * Positivity for CD19+ MRD (molecular failure or molecular relapse), defined as presence of MRD at a level of ≥10^-4 according to an assay with a minimum sensitivity of 10^-4.
   * Donor chimerism <90%, as determined by analysis of host and donor STRs in bone marrow sample engraftment analysis.
3. At least one previous line of treatment for MRD-positivity and/or reduced donor chimerism (i.e. blinatumomab, DLI, TKI or other agents) after allogeneic SCT.
4. For those with BCR/ABL-positive B-precursor ALL only: persistence of MRD and/or MC following at least one ≥ second generation TKI (dasatinib, nilotinib, bosutinib, ponatinib) OR intolerance to second generation TKI and intolerance to or persistence of MRD and/or MC following imatinib mesylate.
5. Availability of allogeneic donor lymphocytes from the subject's donor (at least 2 x 10^8 T cells/kg).
6. Subject has provided written informed consent prior to initiation of any study-specific activities/procedures.
7. Subject has provided informed consent to be followed up in the GMALL-Registry.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.
9. Renal function as follows: serum creatinine < 2.0 mg/dL and estimated glomerular filtration rate > 30 mL/min.
10. Hepatic function as follows:

    * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 3.0 x upper limit of normal (ULN)
    * Alkaline phosphatase (ALP) < 3.0 x ULN
    * Bilirubin ≤ 2.0 x ULN (unless considered due to Gilbert's syndrome or hemolysis)
11. For female subjects only: Women of child-bearing age have to use a reliable method of contraception.

Exclusion Criteria:

1. Eligibility for treatment with blinatumomab ALONE or other antibody-based treatment approaches (e.g. inotuzumab ozogamicin), as considered by the treating physician.
2. Eligibility for standard chemotherapy, as considered by the treating physician.
3. Antitumor therapy (chemotherapy, antibody therapy, molecular-targeted therapy, retinoid therapy, or investigational agent) within 14 days or 5 half-lives (whichever is longer) prior to baseline MRD and/or chimerism assessment.
4. Treatment with systemic immune modulators including, but not limited to, non-topical systemic corticosteroids, cyclosporine, and tacrolimus within 2 weeks before enrollment.
5. Any grade of GvHD currently requiring treatment.
6. Clinically relevant central nervous system (CNS) pathology requiring treatment (e.g., unstable epilepsy).
7. Evidence of current CNS involvement by ALL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of combined DLI and blinatumomab treatment in subjects with treatment-resistant MC or MRD of CD19+ B-precursor ALL after allogeneic SCT | 18 weeks
  Subject incidence and grade of adverse events (AEs) including graft-versus-host disease (GvHD). The intensity of (S)AEs will be assessed according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 4.03.

SECONDARY OUTCOMES:
Efficacy of a combined treatment of DLI and blinatumomab to induce a complete MRD/chimerism response | 18 weeks
  MRD response based on RT-PCR: Complete MRD response (MolCR): hCR and MRD not detectable by molecular probe[s] with a sensitivity ≥10-4. The MRD response is calculated as: [number of patients achieving complete MRD response after at least one cycle (minimum 4 days blinatumomab) of study treatment] / [number of patients who received at least 1 cycle (minimum 4 days blinatumomab) of study treatment].
  Mixed chimerism response: CC response: only donor STRs in bone marrow; Low-level MC response ≥90% but <100% donor STRs in bone marrow. The MC response is calculated as: [number of patients achieving CC/low-level MC response after at least one cycle (minimum 4 days blinatumomab) of study treatment] / [number of patients who received at least 1 cycle (minimum 4 days blinatumomab) of study treatment].
Duration of the response and survival after combined treatment of DLI and blinatumomab | 18 weeks
  For patients who received at least one cycle (minimum 4 days of blinatumomab), progression-free survival and overall survival will be calculated using kaplan-meier survival estimates. Descriptive summary statistics (N, mean, standard deviation, minimum, median and maximum) for the duration of response will be performed for all patients with an observed complete MRD response or CC/low-level MC response.

CONTACTS AND LOCATIONS:
Overall Officials: Marion Subklewe, MD, Principal Investigator — Klinikum der Universität München; Christian Schmidt, MD, Principal Investigator — Klinikum der Universität München; Sascha Haubner, MD, Principal Investigator — Klinikum der Universität München
Locations (1):
- Klinikum der Universität München, Munich, Germany

IPD SHARING:
Plan to Share IPD: Undecided